CLINICAL TRIAL: NCT03430388
Title: Evaluation of Yellow Fever Vaccine in Patients With Rheumatic Diseases Under Low Immunosuppression Level and Residing in a Risk Area
Brief Title: Yellow Fever Vaccine in Patients With Rheumatic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VFAReumatoHC
Record Dates: First submitted 2018-01-30; First posted 2018-02-12 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2018-01

CONDITIONS: Systemic Lupus; Rheumatoid Arthritis; Spondyloarthritis; Inflammatory Myopathy; Systemic Sclerosis; Mixed Connective Tissue Disease; Takayasu Arteritis; Granulomatosis With Polyangiitis; Sjogren's Syndrome; Juvenile Idiopathic Arthritis; Juvenile Dermatomyositis
Keywords: vaccine; Yellow Fever; Rheumatic disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis; Myositis; Scleroderma, Systemic; Mixed Connective Tissue Disease; Takayasu Arteritis; Granulomatosis with Polyangiitis; Sjogren's Syndrome; Arthritis, Juvenile; Dermatomyositis; Yellow Fever; Rheumatic Diseases | interventions — Yellow Fever Vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rheumatic diseases patients (Active Comparator): Vaccination against Yellow Fever, fractional dose (0,1mL) of 17D vaccine
  Interventions: Biological: Yellow Fever vaccine (17D)
- Healthy controls (Active Comparator): Vaccination against Yellow Fever, fractional dose (0,1mL) of 17D vaccine
  Interventions: Biological: Yellow Fever vaccine (17D)

INTERVENTIONS:
Biological: Yellow Fever vaccine (17D) — Vaccination against Yellow Fever, fractional dose (0,1mL) of 17D vaccine

SUMMARY:
According to World Health Organization (WHO), since December 2016, Brazil is showing a significant increase in cases of yellow fever in humans. In view of this, vaccination is suitable for residents and travelers to the risk area. However, for immunosuppressed patients there is a formal recommendation not to vaccinate with live virus vaccine. On the other hand, the safety and efficacy of the vaccine has been demonstrated in patients with HIV, and safety and seroconversion have also been demonstrated in patients with rheumatic disease who were inadvertently revaccinated for yellow fever. Faced with the impossibility of leaving the high-risk area for some patients the vaccination could be released to only those who have low level of immunosuppression as suggested by some recommendations of medical societies. The availability of a fractional vaccine in the State of São Paulo, which has proved its efficacy, opens the possibility of exposure to a lower number of copies of the virus in the first exposure of immunosuppressed patients, allowing, if necessary, a safer revaccination, after 28 days to obtain of a more effective immunogenic response. The objectives of the study are to evaluate the immune response of the immunization with fractional yellow fever vaccine (neutralizing antibodies) in patients with systemic autoimmune rheumatic diseases residing in a high-risk area. Secondarily, evaluate the possible association between immunogenicity and vaccination with: demographic data, clinical and laboratory activity of the disease in patients with chronic rheumatic diseases, evaluate the curve of viremia and report adverse events. Patients and healthy controls will be vaccinated for yellow fever in the Immunization Center of Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (HC-FMUSP). The patients' screening for exclusion and inclusion criteria will be done at the rheumatology outpatient clinic after medical evaluation. For the controls will be the routine screening of the Immunization Center. The vaccination protocol will be a fractional dose of the yellow fever vaccine on day D0 for both groups. Patients will be evaluated on day D0, D5, D10, D30-4 and D365 and controls only on days D0, D10, D30-45 and D365 for aspartate aminotransferase (AST), alanine aminotransferase (ALT), platelets, urea and creatinine, immunoglobulin M (IgM) by immunofluorescence for Yellow Fever, viremia, autoantibodies.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatic disease under low immunosuppression (hydroxychloroquine, sulfasalazine or methotrexate plus prednisone up to 7,5mg/day or leflunomide plus prednisone up to 7,5mg/day),
* Resident in high risk área for Yellow Fever

Exclusion Criteria:

* Active disease
* Primary immunodeficiency
* History of anaphylactic response to vaccine components or egg allergy
* Living outside the risk area
* Do not meet criteria for low immunosuppression
* History of previous immunization with the yellow fever vaccine
* History of live virus vaccine up to 4 weeks before
* Individuals who do not agree to participate in the study and/or whose parents do not agree to participate in the study

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-03-24 (Actual); Study Completion 2019-02-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with severe adverse events to the fractional dose of Yellow Fever vaccine | 10 days
  Comparison of adverse events rates (based on the Brighton Collaboration diagnostic criteria) between rheumatic disease patients and healthy controls after Yellow Fever vaccine
Number of participants with protective levels of antibodies against Yellow Fever vaccine | 30 days
  Comparison of protective antibodies rates (measured by indirect immunofluorescence) against Yellow Fever virus between rheumatic disease patients and healthy controls after Yellow Fever vaccine

SECONDARY OUTCOMES:
Association of number of patients with protective antibodies levels and disease activity in patients with chronic rheumatic diseases | 30 days
  Association of number of patients with protective antibodies levels against yellow fever and disease activity in patients with chronic rheumatic diseases (measured by systemic lupus erythematosus disease activity index-SLEDAI for systemic lupus erythematosus patients, disease activity score-DAS28 for rheumatoid arthritis patients, manual muscle testing-MMT and disease activity score-DAS for inflammatory myopathies patients, Birmingham Vasculitis Activity Score-BVAS for primary vasculitis patients, juvenile arthritis disease activity score-JADAS for juvenile idiopathic arthritis patients)
Number of participants with persistent protective levels of antibodies against Yellow Fever | 1 year
  Comparison of protective antibodies rates (measured by indirect immunofluorescence) against Yellow Fever virus between rheumatic disease patients and healthy controls after Yellow Fever vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Eloisa Bonfa, MD, PhD, Principal Investigator — Rheumatology Division of Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, SP - Brazil
Locations (1):
- Rheumatology Division of Hospital das Clínicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arend WP, Michel BA, Bloch DA, Hunder GG, Calabrese LH, Edworthy SM, Fauci AS, Leavitt RY, Lie JT, Lightfoot RW Jr, et al. The American College of Rheumatology 1990 criteria for the classification of Takayasu arteritis. Arthritis Rheum. 1990 Aug;33(8):1129-34. doi: 10.1002/art.1780330811. PMID 1975175
- [Background] Arnett FC, Edworthy SM, Bloch DA, McShane DJ, Fries JF, Cooper NS, Healey LA, Kaplan SR, Liang MH, Luthra HS, et al. The American Rheumatism Association 1987 revised criteria for the classification of rheumatoid arthritis. Arthritis Rheum. 1988 Mar;31(3):315-24. doi: 10.1002/art.1780310302. PMID 3358796
- [Background] Barte H, Horvath TH, Rutherford GW. Yellow fever vaccine for patients with HIV infection. Cochrane Database Syst Rev. 2014 Jan 23;2014(1):CD010929. doi: 10.1002/14651858.CD010929.pub2. PMID 24453061
- [Background] Bode RK, Klein-Gitelman MS, Miller ML, Lechman TS, Pachman LM. Disease activity score for children with juvenile dermatomyositis: reliability and validity evidence. Arthritis Rheum. 2003 Feb 15;49(1):7-15. doi: 10.1002/art.10924. PMID 12579588
- [Background] Bohan A, Peter JB. Polymyositis and dermatomyositis (first of two parts). N Engl J Med. 1975 Feb 13;292(7):344-7. doi: 10.1056/NEJM197502132920706. No abstract available. PMID 1090839
- [Background] Bombardier C, Gladman DD, Urowitz MB, Caron D, Chang CH. Derivation of the SLEDAI. A disease activity index for lupus patients. The Committee on Prognosis Studies in SLE. Arthritis Rheum. 1992 Jun;35(6):630-40. doi: 10.1002/art.1780350606. PMID 1599520
- [Background] Campi-Azevedo AC, de Almeida Estevam P, Coelho-Dos-Reis JG, Peruhype-Magalhaes V, Villela-Rezende G, Quaresma PF, Maia Mde L, Farias RH, Camacho LA, Freire Mda S, Galler R, Yamamura AM, Almeida LF, Lima SM, Nogueira RM, Silva Sa GR, Hokama DA, de Carvalho R, Freire RA, Filho EP, Leal Mda L, Homma A, Teixeira-Carvalho A, Martins RM, Martins-Filho OA. Subdoses of 17DD yellow fever vaccine elicit equivalent virological/immunological kinetics timeline. BMC Infect Dis. 2014 Jul 15;14:391. doi: 10.1186/1471-2334-14-391. PMID 25022840
- [Background] Cohen JI. Strategies for herpes zoster vaccination of immunocompromised patients. J Infect Dis. 2008 Mar 1;197 Suppl 2(Suppl 2):S237-41. doi: 10.1086/522129. PMID 18419403
- [Background] Consolaro A, Ruperto N, Bazso A, Pistorio A, Magni-Manzoni S, Filocamo G, Malattia C, Viola S, Martini A, Ravelli A; Paediatric Rheumatology International Trials Organisation. Development and validation of a composite disease activity score for juvenile idiopathic arthritis. Arthritis Rheum. 2009 May 15;61(5):658-66. doi: 10.1002/art.24516. PMID 19405003
- [Background] Dougados M, van der Linden S, Juhlin R, Huitfeldt B, Amor B, Calin A, Cats A, Dijkmans B, Olivieri I, Pasero G, et al. The European Spondylarthropathy Study Group preliminary criteria for the classification of spondylarthropathy. Arthritis Rheum. 1991 Oct;34(10):1218-27. doi: 10.1002/art.1780341003. PMID 1930310
- [Background] Esparza RH, Swaak T, Aarden L, Smeenk R. Complement-fixing antibodies to dsDNA detected by the immunofluorescence technique on Crithidia luciliae. A critical appraisal. J Rheumatol. 1985 Dec;12(6):1109-17. PMID 3912506
- [Background] Garrett S, Jenkinson T, Kennedy LG, Whitelock H, Gaisford P, Calin A. A new approach to defining disease status in ankylosing spondylitis: the Bath Ankylosing Spondylitis Disease Activity Index. J Rheumatol. 1994 Dec;21(12):2286-91. PMID 7699630
- [Background] Gladman DD, Ibanez D, Urowitz MB. Systemic lupus erythematosus disease activity index 2000. J Rheumatol. 2002 Feb;29(2):288-91. PMID 11838846
- [Background] Hochberg MC. Updating the American College of Rheumatology revised criteria for the classification of systemic lupus erythematosus. Arthritis Rheum. 1997 Sep;40(9):1725. doi: 10.1002/art.1780400928. No abstract available. PMID 9324032
- [Background] Kuter BJ, Ngai A, Patterson CM, Staehle BO, Cho I, Matthews H, Provost PJ, White CJ. Safety, tolerability, and immunogenicity of two regimens of Oka/Merck varicella vaccine (Varivax) in healthy adolescents and adults. Oka/Merck Varicella Vaccine Study Group. Vaccine. 1995 Aug;13(11):967-72. doi: 10.1016/0264-410x(95)00046-4. PMID 8525689
- [Background] Gershon AA, Steinberg SP. Persistence of immunity to varicella in children with leukemia immunized with live attenuated varicella vaccine. N Engl J Med. 1989 Apr 6;320(14):892-7. doi: 10.1056/NEJM198904063201403. PMID 2538749
- [Background] Leavitt RY, Fauci AS, Bloch DA, Michel BA, Hunder GG, Arend WP, Calabrese LH, Fries JF, Lie JT, Lightfoot RW Jr, et al. The American College of Rheumatology 1990 criteria for the classification of Wegener's granulomatosis. Arthritis Rheum. 1990 Aug;33(8):1101-7. doi: 10.1002/art.1780330807. PMID 2202308
- [Background] Lightfoot RW Jr, Michel BA, Bloch DA, Hunder GG, Zvaifler NJ, McShane DJ, Arend WP, Calabrese LH, Leavitt RY, Lie JT, et al. The American College of Rheumatology 1990 criteria for the classification of polyarteritis nodosa. Arthritis Rheum. 1990 Aug;33(8):1088-93. doi: 10.1002/art.1780330805. PMID 1975174
- [Background] Lovell DJ, Lindsley CB, Rennebohm RM, Ballinger SH, Bowyer SL, Giannini EH, Hicks JE, Levinson JE, Mier R, Pachman LM, Passo MH, Perez MD, Reed AM, Schikler KN, Smith M, Zemel LS, Rider LG. Development of validated disease activity and damage indices for the juvenile idiopathic inflammatory myopathies. II. The Childhood Myositis Assessment Scale (CMAS): a quantitative tool for the evaluation of muscle function. The Juvenile Dermatomyositis Disease Activity Collaborative Study Group. Arthritis Rheum. 1999 Oct;42(10):2213-9. doi: 10.1002/1529-0131(199910)42:103.0.CO;2-8. PMID 10524696
- [Background] Lukas C, Landewe R, Sieper J, Dougados M, Davis J, Braun J, van der Linden S, van der Heijde D; Assessment of SpondyloArthritis international Society. Development of an ASAS-endorsed disease activity score (ASDAS) in patients with ankylosing spondylitis. Ann Rheum Dis. 2009 Jan;68(1):18-24. doi: 10.1136/ard.2008.094870. Epub 2008 Jul 14. PMID 18625618
- [Background] Martins RM, Maia Mde L, Farias RH, Camacho LA, Freire MS, Galler R, Yamamura AM, Almeida LF, Lima SM, Nogueira RM, Sa GR, Hokama DA, de Carvalho R, Freire RA, Pereira Filho E, Leal Mda L, Homma A. 17DD yellow fever vaccine: a double blind, randomized clinical trial of immunogenicity and safety on a dose-response study. Hum Vaccin Immunother. 2013 Apr;9(4):879-88. doi: 10.4161/hv.22982. Epub 2013 Jan 30. PMID 23364472
- [Background] Masi AT, Hunder GG, Lie JT, Michel BA, Bloch DA, Arend WP, Calabrese LH, Edworthy SM, Fauci AS, Leavitt RY, et al. The American College of Rheumatology 1990 criteria for the classification of Churg-Strauss syndrome (allergic granulomatosis and angiitis). Arthritis Rheum. 1990 Aug;33(8):1094-100. doi: 10.1002/art.1780330806. PMID 2202307
- [Background] Moll JM, Wright V. Psoriatic arthritis. Semin Arthritis Rheum. 1973;3(1):55-78. doi: 10.1016/0049-0172(73)90035-8. No abstract available. PMID 4581554
- [Background] Mukhtyar C, Lee R, Brown D, Carruthers D, Dasgupta B, Dubey S, Flossmann O, Hall C, Hollywood J, Jayne D, Jones R, Lanyon P, Muir A, Scott D, Young L, Luqmani RA. Modification and validation of the Birmingham Vasculitis Activity Score (version 3). Ann Rheum Dis. 2009 Dec;68(12):1827-32. doi: 10.1136/ard.2008.101279. Epub 2008 Dec 3. PMID 19054820
- [Background] Oliveira AC, Mota LM, Santos-Neto LL, Simoes M, Martins-Filho OA, Tauil PL. Seroconversion in patients with rheumatic diseases treated with immunomodulators or immunosuppressants, who were inadvertently revaccinated against yellow fever. Arthritis Rheumatol. 2015 Feb;67(2):582-3. doi: 10.1002/art.38960. No abstract available. PMID 25418753
- [Background] Ozen S, Pistorio A, Iusan SM, Bakkaloglu A, Herlin T, Brik R, Buoncompagni A, Lazar C, Bilge I, Uziel Y, Rigante D, Cantarini L, Hilario MO, Silva CA, Alegria M, Norambuena X, Belot A, Berkun Y, Estrella AI, Olivieri AN, Alpigiani MG, Rumba I, Sztajnbok F, Tambic-Bukovac L, Breda L, Al-Mayouf S, Mihaylova D, Chasnyk V, Sengler C, Klein-Gitelman M, Djeddi D, Nuno L, Pruunsild C, Brunner J, Kondi A, Pagava K, Pederzoli S, Martini A, Ruperto N; Paediatric Rheumatology International Trials Organisation (PRINTO). EULAR/PRINTO/PRES criteria for Henoch-Schonlein purpura, childhood polyarteritis nodosa, childhood Wegener granulomatosis and childhood Takayasu arteritis: Ankara 2008. Part II: Final classification criteria. Ann Rheum Dis. 2010 May;69(5):798-806. doi: 10.1136/ard.2009.116657. PMID 20413568
- [Background] Petty RE, Southwood TR, Manners P, Baum J, Glass DN, Goldenberg J, He X, Maldonado-Cocco J, Orozco-Alcala J, Prieur AM, Suarez-Almazor ME, Woo P; International League of Associations for Rheumatology. International League of Associations for Rheumatology classification of juvenile idiopathic arthritis: second revision, Edmonton, 2001. J Rheumatol. 2004 Feb;31(2):390-2. No abstract available. PMID 14760812
- [Background] Prevoo ML, van 't Hof MA, Kuper HH, van Leeuwen MA, van de Putte LB, van Riel PL. Modified disease activity scores that include twenty-eight-joint counts. Development and validation in a prospective longitudinal study of patients with rheumatoid arthritis. Arthritis Rheum. 1995 Jan;38(1):44-8. doi: 10.1002/art.1780380107. PMID 7818570
- [Background] Rider LG, Koziol D, Giannini EH, Jain MS, Smith MR, Whitney-Mahoney K, Feldman BM, Wright SJ, Lindsley CB, Pachman LM, Villalba ML, Lovell DJ, Bowyer SL, Plotz PH, Miller FW, Hicks JE. Validation of manual muscle testing and a subset of eight muscles for adult and juvenile idiopathic inflammatory myopathies. Arthritis Care Res (Hoboken). 2010 Apr;62(4):465-72. doi: 10.1002/acr.20035. PMID 20391500
- [Background] Seror R, Ravaud P, Bowman SJ, Baron G, Tzioufas A, Theander E, Gottenberg JE, Bootsma H, Mariette X, Vitali C; EULAR Sjogren's Task Force. EULAR Sjogren's syndrome disease activity index: development of a consensus systemic disease activity index for primary Sjogren's syndrome. Ann Rheum Dis. 2010 Jun;69(6):1103-9. doi: 10.1136/ard.2009.110619. Epub 2009 Jun 28. PMID 19561361
- [Background] Sidibe M, Yactayo S, Kalle A, Sall AA, Sow S, Ndoutabe M, Perea W, Avokey F, Lewis RF, Veit O. Immunogenicity and safety of yellow fever vaccine among 115 HIV-infected patients after a preventive immunisation campaign in Mali. Trans R Soc Trop Med Hyg. 2012 Jul;106(7):437-44. doi: 10.1016/j.trstmh.2012.04.002. Epub 2012 May 22. PMID 22627101
- [Background] Tanriover MD, Akar S, Turkcapar N, Karadag O, Ertenli I, Kiraz S. Vaccination recommendations for adult patients with rheumatic diseases. Eur J Rheumatol. 2016 Mar;3(1):29-35. doi: 10.5152/eurjrheum.2016.16100. Epub 2015 Oct 28. PMID 27708966
- [Background] van den Hoogen F, Khanna D, Fransen J, Johnson SR, Baron M, Tyndall A, Matucci-Cerinic M, Naden RP, Medsger TA Jr, Carreira PE, Riemekasten G, Clements PJ, Denton CP, Distler O, Allanore Y, Furst DE, Gabrielli A, Mayes MD, van Laar JM, Seibold JR, Czirjak L, Steen VD, Inanc M, Kowal-Bielecka O, Muller-Ladner U, Valentini G, Veale DJ, Vonk MC, Walker UA, Chung L, Collier DH, Csuka ME, Fessler BJ, Guiducci S, Herrick A, Hsu VM, Jimenez S, Kahaleh B, Merkel PA, Sierakowski S, Silver RM, Simms RW, Varga J, Pope JE. 2013 classification criteria for systemic sclerosis: an American College of Rheumatology/European League against Rheumatism collaborative initiative. Arthritis Rheum. 2013 Nov;65(11):2737-47. doi: 10.1002/art.38098. Epub 2013 Oct 3. PMID 24122180
- [Background] van Assen S, Agmon-Levin N, Elkayam O, Cervera R, Doran MF, Dougados M, Emery P, Geborek P, Ioannidis JP, Jayne DR, Kallenberg CG, Muller-Ladner U, Shoenfeld Y, Stojanovich L, Valesini G, Wulffraat NM, Bijl M. EULAR recommendations for vaccination in adult patients with autoimmune inflammatory rheumatic diseases. Ann Rheum Dis. 2011 Mar;70(3):414-22. doi: 10.1136/ard.2010.137216. Epub 2010 Dec 3. PMID 21131643
- [Background] van Assen S, Elkayam O, Agmon-Levin N, Cervera R, Doran MF, Dougados M, Emery P, Geborek P, Ioannidis JP, Jayne DR, Kallenberg CG, Muller-Ladner U, Shoenfeld Y, Stojanovich L, Valesini G, Wulffraat NM, Bijl M. Vaccination in adult patients with auto-immune inflammatory rheumatic diseases: a systematic literature review for the European League Against Rheumatism evidence-based recommendations for vaccination in adult patients with auto-immune inflammatory rheumatic diseases. Autoimmun Rev. 2011 Apr;10(6):341-52. doi: 10.1016/j.autrev.2010.12.003. Epub 2010 Dec 20. PMID 21182987
- [Background] Vitali C, Bombardieri S, Jonsson R, Moutsopoulos HM, Alexander EL, Carsons SE, Daniels TE, Fox PC, Fox RI, Kassan SS, Pillemer SR, Talal N, Weisman MH; European Study Group on Classification Criteria for Sjogren's Syndrome. Classification criteria for Sjogren's syndrome: a revised version of the European criteria proposed by the American-European Consensus Group. Ann Rheum Dis. 2002 Jun;61(6):554-8. doi: 10.1136/ard.61.6.554. PMID 12006334
- [Background] Wu JT, Peak CM, Leung GM, Lipsitch M. Fractional dosing of yellow fever vaccine to extend supply: a modelling study. Lancet. 2016 Dec 10;388(10062):2904-2911. doi: 10.1016/S0140-6736(16)31838-4. Epub 2016 Nov 10. PMID 27837923
- [Derived] Tonacio AC, do Nascimento Pedrosa T, Borba EF, Aikawa NE, Pasoto SG, Filho JCRF, Sampaio Barros MM, Leon EP, Lombardi SCFS, Junior AM, Azevedo AS, Schwarcz WD, Fuller R, Yuki EFN, Ugolini Lopes MR, Rodrigues Pereira RM, Sampaio Barros PD, de Andrade DCO, de Medeiros-Ribeiro AC, de Moraes JCB, Shinjo SK, Miossi R, da Silva Duarte AJ, Lopes MH, Kallas EG, Almeida da Silva CA, Bonfa E. Immunogenicity and safety of primary fractional-dose yellow fever vaccine in autoimmune rheumatic diseases. PLoS Negl Trop Dis. 2021 Nov 29;15(11):e0010002. doi: 10.1371/journal.pntd.0010002. eCollection 2021 Nov. PMID 34843469